CLINICAL TRIAL: NCT02194959
Title: Training African American Peers as Patient Navigators for Colon Cancer Screening
Brief Title: Peer Patient Navigation for Colon Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GCO 07-0594; 5R25CA132692-05 (NIH)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Screening Colonoscopy
Keywords: Patient Navigation; Screening Colonoscopy; Colorectal Cancer Screening; African Americans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peer PN (Experimental): A scheduling phone call will be made to all patients within 14 days of their initial referral to the study. Following the scheduling of their appointment, each patient will be mailed an informational pamphlet with written instructions for the colonoscopy once they have scheduled the procedure. The first reminder PPN phone call will be made two weeks before a patient's scheduled colonoscopy. The second reminder PPN call will be made three days before the scheduled colonoscopy. For all calls, at least three attempts (at different times of the day and different days of the week) will be made to reach patients. All telephone calls will be audio-recorded to facilitate fidelity monitoring. All colonoscopy appointments will be made within the Division of Gastroenterology at each of the hospital sites. The Project Coordinator will be responsible for confirming completion (and no-shows) for all colonoscopy appointments.
  Interventions: Behavioral: Peer PN
- Pro PN (Active Comparator): Participants randomized to standard patient navigation received care that they would normally receive if they were not participating in the study with navigation from the GI staff, and three phone calls that involved scheduling and reminding the participant about their colonoscopy appointment.
  Interventions: Behavioral: Pro PN

INTERVENTIONS:
Behavioral: Peer PN — Navigation by Peer Patient Navigators
  Other Names: Peer Patient Navigation
  Arms: Peer PN
Behavioral: Pro PN — Navigation by Standard Hospital Navigators
  Other Names: Standard Patient Navigation
  Arms: Pro PN

SUMMARY:
Cancer health disparities related to race and ethnicity are among the most serious problems facing the US health care system. A recent institute of medicine report stated that such disparities are seen at every level of health care, from prevention to treatment and follow-up. This problem is acutely evident in the figures for colorectal cancer (CRC) among African Americans. According to the American cancer society, African Americans have the highest CRC incidence and mortality of any ethnic/racial group. Indeed, CRC incidence and mortality are 15% and 43% higher among African Americans than whites, respectively. These disparities could be effectively reduced through greater African American participation in CRC screening and early detection. More importantly, due to the preponderance of CRC in African Americans beyond the reach of the flexible sigmoidoscopy (1), increased adherence to colonoscopy among African Americans will save lives. Although there is clear evidence that providing patients with someone to help them manage/navigate the health care system (i.e., patient navigation (PN)) is effective in helping them to complete cancer screening, very few hospitals provide PN for colonoscopy. The vast majority of hospitals in NYC are unable to provide PN for patients for whom colonoscopy is recommended, in large part because of the costs associated with professional-led PN. This project seeks to address this serious public health problem by investigating the success of training African Americans who have undergone colonoscopy to serve as volunteer peer patient navigators to encourage others from their community to complete CRC screening via colonoscopy.

DETAILED DESCRIPTION:
The overall goal of the study was to reduce CRC morbidity and mortality by increasing African American participation in colonoscopy. This was done by development and implementation of a training program for Peer Patient Navigation (PPN) to increase participation of African Americans in colonoscopy.

The primary care physician referred all participants and introduced the study to the patient. The physician will then introduced the patient to the Research Assistant/Recruiter immediately following the medical visit during which a CRC screening colonoscopy was recommended. The Research Assistant/Recruiter reviewed the study and asked potential participants if they were interested; if so, the candidate's eligibility was determined. If these criteria were met and the patient wanted to be in the study, informed consent and HIPAA was reviewed and obtained. If the patient wanted to think about his/her decision, informed consent was obtained at a later date.

Patients were referred and scheduled for screening colonoscopy as part of standard of care. Both groups received 3 intervention phone calls from their assigned navigators, 1) to schedule the colonoscopy, 2) a call 2 weeks before the procedure and, 3) a third call three days before the procedure.

For research purposes, participants were randomized to one of two kinds of patient navigation:

1. Standard patient navigation receiving care that they would normally receive if they were not participating in the study with navigation from the GI staff, and three phone calls involved scheduling and reminding the participant about their colonoscopy appointment.
2. Peer Patient Navigation (PPN): Participants were assisted by African American peers who have undergone colonoscopy, and were able to discuss, first-hand, their personal experience undergoing colonoscopy and describe how they coped effectively with the procedure.

PPN's underwent three months of training supervised by study investigators. Multiple modes of training were used (didactic discussion, observation, role-playing, one-on-one sessions, ongoing feedback, rehearsal, supervision via review of audio-tape recording or PPNs and a take-home training manual).

A medical chart review was completed after the colonoscopy for all patients to assess completion of the examination as well as prep quality and any findings where additional clinical follow-up was required. Colonoscopy results were also collected to assess quality of care and measure the effectiveness of PPN navigations compared to standard of care, particularly potential differences based on study group, i.e., compliance.

ELIGIBILITY:
Inclusion Criteria:

* Be self-identified as African-American
* Referral from a primary care physician for colonoscopy
* Agree to undergo colonoscopy at a participating hospital
* Be at least 50 years of age or older
* Have telephone service
* Be able to provide informed consent in English

Exclusion Criteria:

* Personal or family history (1st degree relative) of colon cancer
* Personal history of any chronic GI disorder (i.e., irritable bowel syndrome, colitis)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2011-07; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Colonoscopy completion | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lina Jandorf, MA, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Sly JR, Jandorf L, Dhulkifl R, Hall D, Edwards T, Goodman AJ, Maysonet E, Azeez S. Challenges to replicating evidence-based research in real-world settings: training African-American peers as patient navigators for colon cancer screening. J Cancer Educ. 2012 Dec;27(4):680-6. doi: 10.1007/s13187-012-0395-3. PMID 22791543